CLINICAL TRIAL: NCT05109962
Title: New Recommendations for Robertsonian Translocation Management After Preimplantation Genetic Testing of Structural Rearrangement (PGT-SR) Attempts: What Should be Done With Mosaic Embryos?
Brief Title: Management of Robertsonian Translocation PGT-SR Attempts
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0452
Record Dates: First submitted 2021-07-05; First posted 2021-11-05 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-10

CONDITIONS: Robertsonian Translocation
Keywords: Several years of miscarriages; Abortions and primary infertility; FISH with 2 probes; FISH with 3 probes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — NC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
to analyze if a probe strategy choice for PGT-SR studies of Robertsonian translocations (RT) influences the fate of embryos? Few studies discussed the importance of probe choices. However, those who did, demonstrated that analysis with locus specific probes improve a diagnosis of dubious results, and addition of a centromeric probe could affect the accuracy of diagnosis

ELIGIBILITY:
Inclusion criteria:

* Adult patient whom carrying robertsonian translocations in the context of PGT-SR management
* age > 18 years

Exclusion criteria:

- age < 18 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Robertsonian translocation carriers are phenotypically normal, but they are known to be at increased risk of repeated miscarriages compared with the general population estimated at about 15% of pregnancies, and also resulting in the birth of a child with congenital anomalies or a mental retardation.
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants with detect all chromosome segments | 1 day
  Number of Participants with detect all chromosome segments

CONTACTS AND LOCATIONS:
Overall Officials: Reda Zenagui, PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC